CLINICAL TRIAL: NCT06409117
Title: 3rd Generation Resorbable Magnesium Scaffolds vs Biodegradable Polymer Drug Eluting Stents in Patients With Non ST-segment Elevation Acute Coronary Syndromes: the RESORB-ACS Randomized Clinical Trial
Brief Title: 3rd Generation Resorbable Magnesium Scaffolds vs Biodegradable Polymer Stents in NSTE/ACS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Konstantinos Toutouzas (Other)
Collaborators: Centre Hospitalier Universitaire Saint Pierre (Other); Université Catholique de Louvain (Other); University Hospital of Leuven Leuven (Other); University of Patras (Other); Ippokrateio General Hospital of Thessaloniki (Other)
Responsible Party: Sponsor-Investigator, Konstantinos Toutouzas, Professor of Cardiology, National and Kapodistrian University of Athens
Organization: National and Kapodistrian University of Athens (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESORB-ACS
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Acute Coronary Syndrome; Coronary Artery Disease
Keywords: PCI; NSTE/ACS; resorbable magnesium scaffolds; Scaffolds
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: 3rd generation resorbable magnesium scaffolds "Freesolve" will be compared to the biodegradable polymer drug eluting stents "Orsiro" in patients with NSTE/ACS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resorbable magnesium scaffold (Active Comparator): 3rd generation resorbable magnesium scaffolds
  Interventions: Device: Percutaneous coronary intervention
- Drug eluting stent (Active Comparator): Biodegradable polymer drug eluting stents
  Interventions: Device: Percutaneous coronary intervention

INTERVENTIONS:
Device: Percutaneous coronary intervention — Percutaneous coronary intervention with scaffold implantation in patients with NSTE/ACS

SUMMARY:
This is a multicentre, prospective, randomized controlled trial that will investigate the role and performance of the 3rd generation resorbable magnesium scaffolds "DREAMS 3G" labeled under the name "Freesolve" vs contemporary biodegradable polymer scaffolds in non ST-segment elevation acute coronary syndromes. Patients fulfilling the eligibility criteria will be enrolled and undergo PCI with either Freesolve or Orsiro platforms for the culprit lesion only. They will be followed-up for 12 months (1, 6 and 12 months). The primary endopoint will be Target Lesion Failure as defined by ARC definitions.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE Scaffolding the coronary vessels while maintaining the physiological and rheological properties was an appealing idea resulting in the development of the bioresorbable scaffolds (BRS). The most thoroughly studied BRS - the poly-L-lactide acid based BRS ABSORB™ - evidenced increased rates of device-related adverse events in the randomized controlled trials (RCT) and was removed from market in 2017. ABSORB was an everolimus eluting BRS, characterized by limited radial force, thicker and wider struts, unfavorable crossing profile and unpredictable resorption.

In an effort to overcome these obstacles, metallic resorbable scaffolds were developed - with the main representative being the resorbable magnesium scaffolds (RMS). The absorbable metal stent (AMS) (BIOTRONIK AG, Bülach, Switzerland). was the first device tested in the PROGRESS-AMS trial showing feasibility but necessity for improvement. DREAMS 1G (BIOTRONIK AG, Bülach, Switzerland) was the first generation of the improved RMS, designed to improve radial force and coated with a paclitaxel-polymer matrix. It was studied in the BIOSOLVE-I and showed improved performance compared to the AMS with no probable or definite scaffold thrombosis, however late-lumen-loss (LLL) was relatively high compared to ABSORB scaffolds and contemporary drug eluting stents (DES).

The second generation was the DREAMS 2G (BIOTRONIK AG, Bülach, Switzerland), gaining CE-Mark in 2016 and marketed as Magmaris™. It is designed with more flexible and stronger scaffold backbone targeting in improved radial force with 150x140μm strut thickness. The drug-polymer coating was substituted by the sirolimus BIOlute™ matrix of the Orsiro™ DES, to decrease more effectively neointimal formation. Also, radiopaque markers were added for enhanced x-ray visibility. The outcomes of Magmaris™ have been investigated in the BIOSOLVE II, III, IV trials. In summary, BIOSOLVE II and III demonstrated no scaffold thrombosis with improved LLL improved to its precursor and BIOSOLVE IV exhibited low event rates in a large single-arm study.

The concept of protecting the vulnerable, eroded or ruptured plaque without a permanent metallic endoprosthesis finds ideal application in the acute coronary syndromes. Culprit lesions present as a ruptured plaque, plaque erosion or less frequently as a calcific nodule complicated by thrombotic burden and implantation of a BRS may adequately revascularize the vessel, protect the lesion and be resorbed after vessel healing restoring its elastic and hydraulic properties. However, the high thrombotic status of an acute coronary syndrome (ACS) was preventing BRS of being utilized in such situations. The TROFI-II RCT compared the ABSORB scaffold with DES in ST-segment elevation myocardial infarction (STEMI) and 6-month results were comparable. The Magmaris™ was tested in STEMI patients in the MAGSTEMI RCT and showed significantly higher vasodilatory response at 1-year compared to Orsiro™. Furthermore, Magmaris™ did not raise thrombotic concerns, but resulted in higher target lesion revascularization (TLR) rates although not powered for those endpoints. The BESTMAG trial was a small propensity-matching study providing hypothesis generating outcomes of numerically higher TLR rates with Magmaris™ compared to contemporary biodegradable polymer (BP) or durable polymer (DP)-DES in STEMI presentations. The BIOSOLVE IV registry (n=206) underwent PCI because of non ST-segment elevation (NSTE) myocardial infarction and target vessel failure (TVL) was calculated at 6.1% in 12 months. One death (0.5%) and 2 thrombotic complications were reported (1%). Smaller registries that included NSTE/ACS patients treated with Magmaris™ RMS demonstrated zero deaths and scaffold thrombosis, albeit these are hypothesis generating results limited by the small sample.

The BIOMAG-I first-in-human study investigated the third generation Freesolve™ RMS. The main characteristics are a refined magnesium alloy to enhance scaffolding properties, increased scaffold marker x-ray visibility, larger size range, thinner strut thickness and predictable full resorption in about 12 months. The 1-year results of the BIOMAG-I showed lower LLL (38% lower) than the BIOSOLVE II, low target lesion failure (TLF) rates and no death, target vessel myocardial infarction (MI) or scaffold thrombosis. Of note no struts ware visible in the 1-year optical coherence tomography (OCT). 20.7% of the patients presented with NSTE myocardial infarction lesions and were treated accordingly.

The current guidelines of the European Society of Cardiology recommend use of the BRS only in the context of clinical trials. However, more data and devices are available to hypothesize that RMS may provide a potentially reliable and safe alternative to DES. This trial will further investigate and evaluate the safety and efficacy of the 3rd generation Freesolve™ RMS in NSTE/ACS patients.

STUDY PROCEDURES Screening Patients who will undergo coronary angiography because of NSTE/ACS will be screened for eligibility criteria after signing the informed consent. Demographics, medical history, clinical examination, 12-lead electrocardiogram and per local practice blood laboratory tests will be performed. For women of child-bearing potential, a blood pregnancy test must be performed.

Randomization - enrolment Patients screened and fulfilling eligibility criteria will be enrolled after signing the informed consent form as per RESORB-ACS enrolment and follow-up algorithms (Figure 1). They will be randomly assigned in 1:1 ratio to receive either the Freesolve™ RMS or the BP DES Orsiro® for the PCI of the index NSTE/ACS culprit vessel. The Intention to Treat (ITT) and the Per Protocol (PP) population will only be based on enrolled subjects.

Index PCI All patients enrolled will undergo PCI of the culprit lesion according on the local practice. The instruction for use (IFU) will be followed for every scaffold implantation. In the BP DES arm, the standard DES PCI procedure per local practice will be followed.

Post-procedural care Patients enrolled that have undergone PCI will receive standard NSTE/ACS and post-PCI care in each centre. Double antiplatelet treatment is recommended for at least 12 months.

Follow-up Follow-up will be performed at 1, 6, 12 months and annually up to 36 months follow-up. (visit window ± 10 days). In case that there is no adverse event or complaint from the patient that requires physical examination, the follow-up visits may be conducted through telephone or video call with the investigators.

Study exit Screen failure, withdrawal of the informed consent, lost to follow-up and PCI without scaffold implantation will result in early termination.

Study completion Subject who completes all protocol-required study procedures and follow-ups will complete the trial.

Examinations Clinical examination including angina status or myocardial ischemia, 12-lead electrocardiogram and per local practice blood laboratory tests including will be performed at screening, and during hospitalization post-PCI. Follow-ups will be clinically driven with thorough history primarily focused on any possible myocardial ischemia symptoms. Based on the investigators' - treating physicians' clinical suspicion more examination may be performed to investigate the existence of adverse events/endpoints.

PROCEDURAL DETAILS The device The Freesolve™ scaffold is a Magnesium alloy fully resorbable scaffold developed by BIOTRONIC and represents the 3rd generation of RMS (DREAMS 3G). It is indicated for improving the luminal diameter for treatment of de novo coronary artery lesions by PCI.

Freesolve™ is a scaffold system consisting of a balloon-expandable bioabsorbable scaffold pre-mounted on the balloon of a rapid-exchange PTCA catheter. The scaffold backbone is made from bioabsorbable Magnesium and contains two permanent x-ray markers made from Tantalum on the distal and on the proximal scaffold end, respectively. The surface of the scaffold backbone is completely coated with bioresorbable PLLA (Poly-L-Lactidic Acid) which incorporates Sirolimus. Sirolimus load is 1.4 ± 0.3 μg per mm2 scaffold surface. The DREAMS 3G scaffold system is packaged in a dispenser. The dispenser is placed in an aluminium Tyvek pouch. The device is sterilized using ethylene oxide sterilization. In vivo investigations using a porcine model show that DREAMS 3G provides vessel support for about 3-6 months and releases around 70% Sirolimus from the PLLA carrier during a period of 3 months after implantation. The drug coating is based on the BIOlute® platform.

Training The operators and the operating teams that are going to participate in this protocol and implant the RMS have to be trained on the consensus paper by Fajadet et al. and follow the "4P" principles.

Device implantation - procedure The RMS Freesolve™ is available in 2.5mm, 3mm, 3.5mm and 4mm diameter and in 13mm, 22mm length for all diameters and 26mm/30mm length for the 3mm, 3.5 mm and 4mm diameters. It can be expander after post-dilatation up to 0.6mm in diameter. Nominal pressure for implantation inflation is 10atm and rated burst pressure 16atm. It is delivered through 6Fr guiding catheter and over angioplasty 0.014'' wires.

Following intracoronary injection of nitroglycerin or isosorbide dinitrate, a baseline angiography of the target vessel must be performed in at least 2 orthogonal views, presenting the target lesion free of foreshortening or vessel overlap. In addition to the clinical routine, OCT and intravascular ultrasound (IVUS) documentation may be done pre-PCI per operator's discretion. By intravascular imaging, detailed examination of the lesion as well as accurate length and reference diameter can be performed.

Lesion access is up to the discretion of the investigator. Pre-dilatation of the target lesion is mandatory. The use of intravascular lithotripsy, drug coated balloons or rotational/orbital atherectomy device is not allowed. Pre-dilatation with a non-compliant balloon with a 1:1 balloon-to-artery ratio is mandatory. The balloon should expand fully with no "waist" at full expansion. Non-compliant balloons are more predictable and are recommended. The residual stenosis before the RMS implantation is required to be ≤ 20%, confirmed by any method and TIMI flow should be III.

The scaffold length should cover the target lesion from normal reference vessel diameter proximally to normal vessel distally to assure full coverage of the lesion. The diameter of the RMS should be chosen as following: 2.5mm for 2.5-2.7mm distal reference diameter (DRD), 3.0mm for 2.7-3.2mm DRD, 3.5mm for 3.2-3.7mm DRD, 4.0mm for 3.7-4.2 DRD. The length should be chosen based on the lesion length by angiography or IVUS, OCT. Only one clinical investigation scaffold should be used per lesion. After scaffold implantation an angiography must be performed following intracoronary injection of nitroglycerine or isosorbide dinitrate. Post-dilatation with a non-compliant balloon of up to 0.5 mm larger than the nominal scaffold size and at high pressure (>16 atm) is mandatory. The use of cutting/scoring or drug coated balloons after RMS implantation is not allowed. After post-dilatation, all subjects will undergo the routine angiography and possibly OCT/IVUS. Intravascular imaging may evaluate expansion, apposition and any possible edge or in-scaffold complication.

Culprit lesion In NSTE/ACS identification of the culprit lesion might be challenging. Investigational data with cardiac magnetic resonance imaging identification has showed that in up to 27% of the NSTE/ACS patients' revascularization has been performed in non-culprit lesions. Moreover, electrocardiographic identification is neither sensitive nor specific and recent data demonstrated that in 14% of the studied patients, conventional angiography failed to identify the culprit lesion. In those ambiguous cases, intravascular imaging with IVUS or OCT plays a critical role in the characterization and identification of the culprit lesion. In the RESORB-ACS trial, operators will decide about the possible culprit lesion and that decision may be assisted and guided by intravascular imaging in case it is needed.

Multivessel disease Multivessel disease is not an exclusion criterion except for the cases that CABG is programmed. Enrolled subjects may undergo PCI with RMS only for the culprit lesion during the index procedure. However, in cases that multivessel disease amenable to PCI is present, operators can proceed to full revascularization with conservative DES or Freesolve™ RMS.

Treatment failure and bailout situation For dissections occurring during, or immediately after implantation of RMS, a second RMS may be used, not overlapping with initial one but implanted end-to- end. If another stent needs to be implanted in the immediate vicinity of an already implanted RMS only a Freesolve™ coronary scaffold system should be used. Contact of the Freesolve™ with an uncoated or polymer coated stent up to 120 days may result in accelerated resorption of the DREAMS 3G and undesired local and downstream effects. After 120 days any other stent type may be used. In case of bailout, If a Freesolve™ is not possible to be used, an Orsiro® DES with its proBIO® passive coating and BIOlute® active coating is recommended to be implanted directly adjacent or minimally overlapping based on the consensus recommendations.

Medication Every patient included in this trial must be able to receive 12-month DAPT with aspirin and clopidogrel or ticagrelor or prasugrel. The timing and necessity (in case the patient was already under antiplatelet treatment) will be at the discretion of the treating physician. At all cases DAPT must be present at the time of the implantation based on the ESC guidelines doses for the management of ACS. The use of anticoagulation during PCI (heparin or enoxaparine) at therapeutic dose for PCI will be chosen by the operators. IIb/IIIa glycoprotein inhibitors as well as vasomotor medications will be left at operators' discretion. After the PCI, all patients must receive at least 12-month DAPT. After 12 months, DAPT may be changed to single treatment with aspirin/clopidogrel/ticagrelor/prasugrel or prolonged based on the balance of ischemic/hemorrhagic risk of the patient. Regarding patients receiving oral anticoagulation (eg atrial fibrillation, prosthetic valve, thrombophilia) we recommend that DAPT should be maintained until 1-month follow-up. Afterwards DAPT can be downsized to either aspirin or clopidogrel alone combined with oral anticoagulant for the remaining time period up to 12 months. After 12 months, monotherapy with oral anticoagulant may be prescribed and continued indefinitely.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years old.
2. Patient understands the purpose, the potential risks as well as benefits of the trial and is willing to participate in all parts of the follow-up.
3. Patient has given written consent to participate in the trial.
4. Patients presenting with NSTE/ACS documented in an emergency department or cath lab fulfilling the NSTE/ACS definition of the ESC guidelines (18, 20).
5. Patients undergoing PCI for the index NSTE/ACS.
6. Reference index vessel diameter between 2.5-4.2 mm and length ≤28mm by visual estimation.
7. Lesion preparation by either manual thrombectomy or pre-dilatation has been successful, with opening of the vessel and Thrombolysis in Myocardial Infarction (TIMI) flow >2 and residual stenosis <20%.
8. Culprit lesion treatment only in the index procedure with planned implantation of one only RMS.
9. Patients who have no contraindication for.dual antiplatelet therapy (DAPT).

Exclusion Criteria:

1. A known hypersensitivity or contraindication to any of the following: aspirin, heparin, ticagrelor, prasugrel, bivalirudin, clopidogrel, scaffold material, contrast media, sirolimus.
2. Ongoing infection, including active endocarditis.
3. NSTE/ACS due to in stent/scaffold thrombosis/restenosis.
4. Severely tortuous, angulated or calcified coronary arteries resulting in not successful pre-dilatation or complication as described in exclusion criteria 10.
5. Culprit vessel left main.
6. Ostial target lesion (within 5.0 mm of vessel origin).
7. Bifurcation target lesions Medina 1,1,1 with upfront planned 2-stent technique.
8. Bifurcation side branch target lesions Medina 0,0,1.
9. Known thrombocytopenia (PLT<100,000/mm3).
10. Unsuccessful pre-dilatation, defined as a residual stenosis rate more than 20%, estimated by any method and/or angiographic complications (e.g. distal embolization, side branch closure, extensive dissections).
11. Culprit lesion requiring preparation with technique other than semi/non-compliant and/or cutting/scoring balloons (eg rotational/orbital atherectomy, shockwave lithotripsy).
12. Planned PCI in more lesions than the culprit one at the index procedure.
13. Culprit vessel located or supplied by bypass graft.
14. Life expectancy less than 1 year.
15. Active severe bleeding (Bleeding Academic Research Consortium classification ≥III) (21).
16. Cardiogenic shock.
17. Major surgery planned into the next 6 months that requires double antiplatelet treatment discontinuation.
18. Diffuse severe coronary artery disease that will require coronary artery bypass grafting (CABG) planned in the next 6 months.
19. Chronic kidney disease with eGFR<15 ml/min or under dialysis.
20. Enrolment in another study that competes or interferes with this study.
21. Subject will not be able to comply with the follow-up requirements according to investigators' opinion.
22. Pregnant or breast-feeding females or females who intend to become pregnant during the time of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure rates | 12 months
  cardiovascular death, myocardial infarction (target vessel) and target lesion renascularization (clinically driven)

SECONDARY OUTCOMES:
Target lesion revascularization rates | 1, 6, 12 months and annually up to 36 months
  Clinically driven target lesion revascularization
Cardiac death rates | 1, 6, 12 months and annually up to 36 months
  Cardiac death
All-cause mortality rates | 1, 6, 12 months and annually up to 36 months
  All-cause mortality
Target vessel myocardial infarction rates | 1, 6, 12 months and annually up to 36 months
  Target vessel myocardial infarction
Definite and probable scaffold thrombosis rates | 1, 6, 12 months and annually up to 36 months
  Definite and probable scaffold thrombosis
Device success rates | Peri-procedurally
  Device success defined as final residual diameter stenosis of <30% by angiographic visual assessment using the assigned device only and successful delivery of the RMS/DES to the target lesion, appropriate RMS/DES deployment, successful removal of the delivery system.

CONTACTS AND LOCATIONS:
Overall Officials: Leonidas Koliastasis, MD, PhD, Study Director — National and Kapodistrian University of Athens, CHU Saint-Pierre; Konstantinos Toutouzas, Professor, Principal Investigator — National and Kapodistrian University of Athens; Quentin de Hemptinne, Professor, Principal Investigator — Centre Hospitalier Universitaire Saint Pierre
Locations (7):
- Belgium (4):
  - CHU Saint-Pierre, Brussels
  - UZ Brussel, Brussels
  - UZ Leuven, Leuven
  - UC Louvain, Leuven
- Greece (2):
  - Hippocration Hospital, Athens, Attica
  - Hippokration hospital, Thessaloniki
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Haude M, Wlodarczak A, van der Schaaf RJ, Torzewski J, Ferdinande B, Escaned J, Iglesias JF, Bennett J, Toth GG, Joner M, Toelg R, Wiemer M, Olivecrano G, Vermeersch P, Garcia-Garcia HM, Waksman R. A new resorbable magnesium scaffold for de novo coronary lesions (DREAMS 3): one-year results of the BIOMAG-I first-in-human study. EuroIntervention. 2023 Aug 7;19(5):e414-e422. doi: 10.4244/EIJ-D-23-00326. PMID 37334655
- [Result] Verheye S, Wlodarczak A, Montorsi P, Torzewski J, Bennett J, Haude M, Starmer G, Buck T, Wiemer M, Nuruddin AAB, Yan BP, Lee MK. BIOSOLVE-IV-registry: Safety and performance of the Magmaris scaffold: 12-month outcomes of the first cohort of 1,075 patients. Catheter Cardiovasc Interv. 2021 Jul 1;98(1):E1-E8. doi: 10.1002/ccd.29260. Epub 2020 Sep 3. PMID 32881396
- [Result] de Hemptinne Q, Xaplanteris P, Guedes A, Demeure F, Vandeloo B, Dugauquier C, Picard F, Warne DW, Pilgrim T, Iglesias JF, Bennett J. Magmaris Resorbable Magnesium Scaffold Versus Conventional Drug-Eluting Stent in ST-Segment Elevation Myocardial Infarction: 1-Year Results of a Propensity-Score-Matching Comparison. Cardiovasc Revasc Med. 2022 Oct;43:28-35. doi: 10.1016/j.carrev.2022.05.028. Epub 2022 May 26. PMID 35641364
- [Result] Koliastasis L, Bennett J, Xaplanteris P, Skalidis I, Guedes A, Demeure F, Vandeloo B, Dugauquier C, Picard F, Warne DW, Pilgrim T, Iglesias JF, de Hemptinne Q. Two-year clinical outcomes of resorbable magnesium scaffold versus conventional drug-eluting stents in ST-segment elevation myocardial infarction: A propensity score matching analysis. Hellenic J Cardiol. 2024 Jul-Aug;78:84-86. doi: 10.1016/j.hjc.2023.12.004. Epub 2023 Dec 21. No abstract available. PMID 38134970
- [Result] Sabate M, Alfonso F, Cequier A, Romani S, Bordes P, Serra A, Iniguez A, Salinas P, Garcia Del Blanco B, Goicolea J, Hernandez-Antolin R, Cuesta J, Gomez-Hospital JA, Ortega-Paz L, Gomez-Lara J, Brugaletta S. Magnesium-Based Resorbable Scaffold Versus Permanent Metallic Sirolimus-Eluting Stent in Patients With ST-Segment Elevation Myocardial Infarction: The MAGSTEMI Randomized Clinical Trial. Circulation. 2019 Dec 3;140(23):1904-1916. doi: 10.1161/CIRCULATIONAHA.119.043467. Epub 2019 Sep 25. PMID 31553204
- [Result] Fajadet J, Haude M, Joner M, Koolen J, Lee M, Tolg R, Waksman R. Magmaris preliminary recommendation upon commercial launch: a consensus from the expert panel on 14 April 2016. EuroIntervention. 2016 Sep 18;12(7):828-33. doi: 10.4244/EIJV12I7A137. PMID 27639734